CLINICAL TRIAL: NCT04331639
Title: Implementation of High Dose Interval Vitamin D Supplementation in Patients With Inflammatory Bowel Disease Receiving Infliximab or Vedolizumab
Brief Title: High Dose Interval Vitamin D Supplementation in Patients With Inflammatory Bowel Disease Receiving Biologic Therapy
Status: Recruiting | Type: Observational
Sponsor: Boston Children's Hospital (Other)
Responsible Party: Principal Investigator, Rebecca Gordon, Attending Physician, Boston Children's Hospital
Other Study IDs: P00033424
Record Dates: First submitted 2020-03-23; First posted 2020-04-02 (Actual); Last update posted 2025-03-03 (Actual); Status verified 2025-02

CONDITIONS: Inflammatory Bowel Disease; Crohn Disease; Ulcerative Colitis; Vitamin D Deficiency
MeSH Terms: conditions — Inflammatory Bowel Diseases; Crohn Disease; Colitis, Ulcerative; Vitamin D Deficiency | interventions — Cholecalciferol

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Dietary Supplement: vitamin D3 — Subjects will receive oral high dose interval vitamin D3, concurrently when they are receiving their biologic treatment for their inflammatory bowel disease every 4-8 weeks.
  Other Names: cholecalciferol

SUMMARY:
The investigators will be administering oral high dose interval vitamin D, concurrently when participants are receiving biologic therapy for their inflammatory bowel disease. The investigators will be collecting some additional bloodwork and questionnaires at the time of participants infusions.

DETAILED DESCRIPTION:
The investigators will be administering oral high dose interval vitamin D3 concurrently when participants with inflammatory bowel disease (IBD) are receiving biologic therapy every 4-8 weeks. The investigators will collect additional bloodwork when participants are getting clinical labwork in order to assess markers of bone health and inflammation in response to vitamin D treatment. The investigators will serially assess with questionnaires associated measures, including dietary vitamin D and calcium intake, sunlight exposure, physical activity, fracture history, IBD disease activity, and overall health.

ELIGIBILITY:
Inclusion Criteria:

* Existing diagnosis of IBD, including Crohn disease, ulcerative colitis, and indeterminate colitis
* Receiving treatment with Infliximab or Vedolizumab every 4-8 weeks
* Age 5-25 years old, at study entry
* Measured serum level of 25-OHD of less than 40 ng/mL in the last 4-8 weeks and no changes in vitamin D supplementation in the interim. Of note, 25-OHD levels are evaluated routinely as part of standard clinical care for IBD

Exclusion Criteria:

* History of any underlying kidney disease
* History of preexisting liver disease
* History of granulomatous disease
* Inability to take oral vitamin D3 as a pill
* History of hypercalcemia or hypercalciuria
* Currently, or within the past 3 months, taking an anti-epileptic medication or Lasix

Ages: 5 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Gender Based: Yes
Study Population: See above. Enrolling all eligible participants, who wish to participate, until reach enrollment target.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2020-11-01 (Actual); Primary Completion 2024-09-01 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
vitamin D target | at study conclusion, up to 64 weeks
  assessment of the percentage of patients achieving a serum 25-OHD level in the range of 40-60 ng/mL

SECONDARY OUTCOMES:
change in vitamin D level | at study conclusion, up to 64 weeks
  assess change in serum 25-OHD level from study entry to study conclusion
vitamin D binding protein | at between 12 and 24 weeks (midway through study) and up to 64 weeks (at study conclusion)
  assessing vitamin D binding protein and free vitamin D
parathyroid hormone | at between 12 and 24 weeks (midway through study) and up to 64 weeks (at study conclusion)
  assessing parathyroid hormone
serum safety parameter | at between 12 and 24 weeks (midway through study) and up to 64 weeks (at study conclusion)
  evaluate serum calcium level
urine safety parameter | at between 12 and 24 weeks (midway through study) and up to 64 weeks (at study conclusion)
  evaluate urinary calcium to creatinine ratio
bone mineral density | at study conclusion, up to 64 weeks, when clinically available
  assess changes in bone density and body composition as assessed by DXA scan, when clinically available
markers of bone turnover | at between 12 and 24 weeks (midway through study) and up to 64 weeks (at study conclusion)
  evaluating bone turnover markers such as c-telopeptide, bone specific alkaline phosphatase, osteocalcin, and N-terminal propeptide of type 1 procollagen. May do some of these, and then depending upon the results, consider doing additional analytes, as exploratory analysis.
inflammatory bowel disease treatment parameters | at between 12 and 24 weeks (midway through study) and up to 64 weeks (at study conclusion)
  assess level of Inflixmab, including antibodies to Infliximab and Infliximab levels, when clinically available
cytokine measurements | at 0 weeks (entry into study) and up to 64 weeks (at study conclusion)
  evaluating pro-inflammatory and anti-inflammatory cytokine levels, specifically interleukin-17 and interferon gamma, with likely additional exploratory studies to further characterize immune response to vitamin D repletion depending upon these results.
c-reactive protein | at all study time points, from 0 weeks (entry into study) to up to 64 weeks (at study conclusion), as clinically available
  evaluating c-reactive protein
erythrocyte sedimentation rate | at all study time points, from 0 weeks (entry into study) to up to 64 weeks (at study conclusion), as clinically available
  evaluating erythrocyte sedimentation rate
health-related quality of life questionnaire for inflammatory bowel disease | at 0 weeks (entry into study) and up to 64 weeks (at study conclusion)
  assess quality of life measures in children with inflammatory bowel disease
baseline questionnaire on overall health | at 0 weeks (entry into study)
  assess overall health questionnaire
fracture history questionnaire | at 0 weeks (entry into study)
  assess fracture history
food frequency questionnaire | at 0 weeks (entry into study)
  assess calcium and vitamin D food frequency
physical activity questionnaire | at 0 weeks (entry into study) and up to 64 weeks (at study conclusion)
  assess physical activity level
sun exposure questionnaire | at 0 weeks (entry into study) and up to 64 weeks (at study conclusion)
  assess sunlight exposure
follow-up questionnaire on overall health | at 4 weeks to up to 64 weeks, at all study visits except the initial visit (0 weeks)
  assess for any changes in inflammatory bowel disease treatment since last visit

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca Gordon, MD, Principal Investigator — Boston Children's Hospital
Locations (1):
- Boston Children's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No